CLINICAL TRIAL: NCT04030143
Title: A Phase 1b, Open-label, Multiple-dose, Randomized, Parallel-arm, Safety, Tolerability, and Pharmacokinetic Trial of Aripiprazole Intramuscular Depot Administered in the Gluteal Muscle in Adult Subjects With Schizophrenia or Bipolar I Disorder
Brief Title: A Trial of Multiple-doses of Aripiprazole in Adults With Schizophrenia or Bipolar 1 Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 031-201-00181
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia; Bipolar I Disorder
Keywords: Aripiprazole; Aripiprazole Intramuscular Depot; Gluteal Muscle; Long Acting Injection
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder (Experimental): Participants with schizophrenia or bipolar I disorder received aripiprazole 2 month (2M) long-acting injection (LAI) 960 milligrams (mg) for a total of 4 injections administered every 56 days (± 2 days) over the course of 32 weeks.
  Interventions: Drug: Aripiprazole
- Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder (Experimental): Participants with schizophrenia or bipolar I disorder received aripiprazole IM 400 mg, for a total of 8 injections administered every 28 days (± 2 days) over the course of 32 weeks.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Administered as an intramuscular (IM) depot injection.
  Other Names: OPC-14597; Lu AF41155
  Arms: Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Drug: Aripiprazole — Administered as an IM depot injection.
  Other Names: OPC-14597; Lu AF41155
  Arms: Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder

SUMMARY:
The purpose of this trial is to determine the safety and tolerability of multiple-dose administrations of aripiprazole, to establish the similarity of aripiprazole concentrations on the last day of the dosing interval following the final administration of aripiprazole into the gluteal muscle site, and to establish the similarity of aripiprazole exposure over the dosing interval following the administration of aripiprazole into the gluteal muscle site in adult participants with schizophrenia or bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* A current diagnosis of schizophrenia or bipolar I disorder, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
* Body mass index of 18 to 35 kilograms per meter square (kg/m^2).
* On a stable dose of an atypical oral antipsychotic medication for at least 2 months prior to screening.

Exclusion Criteria:

* Participants who have:

  * Met DSM-5 criteria for substance use disorder within the past 180 days.
  * A positive drug screen for drugs of abuse
* Use of any psychotropic medications other than their current non-aripiprazole antipsychotic or mood stabilizer(s) medication; or participants who use more than one antipsychotic or mood stabilizer(s) medication at screening.
* Females who are pregnant, breast-feeding, lactating, and/or have a positive pregnancy test result prior to receiving investigational medicinal product (IMP). A negative serum pregnancy test must be confirmed prior to the first dose of IMP for all female participants.
* Any major surgery within 30 days prior to enrollment or scheduled/elective surgery during the trial.
* Evidence of organ dysfunction or any clinically significant deviation from normal in the physical, electrocardiographic, or clinical laboratory examinations.
* Participants currently in an acute relapse of schizophrenia.
* Participants with a current DSM-5 diagnosis other than schizophrenia or bipolar I disorder, including schizoaffective disorder, major depressive disorder, delirium, dementia, amnestic, or other cognitive disorders. Also, participants with borderline, paranoid, histrionic, or antisocial personality disorder.
* Participants with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia.
* History of any significant drug allergy or known or suspected hypersensitivity, in particular to aripiprazole or other quinolinones.
* History of or current hepatitis or acquired immunodeficiency syndrome or carriers of Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies (anti-HCV), and/or Human immunodeficiency virus (HIV) antibodies.
* Participants deemed intolerant of receiving injections.
* Participants who have had electroconvulsive therapy within 2 months of administration of IMP.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 266 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland International Research Group, Rogers, Arkansas
  - CITrials - Bellflower, Bellflower, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - California Clinical Trials Medical Group, Glendale, California
  - Synergy Research Centers, Lemon Grove, California
  - NRC Research Institute, Orange, California
  - California Neuropsychopharmacology Clinical Research Institute San Diego, San Diego, California
  - Collaborative Neuroscience Network - South Bay, Torrance, California
  - Research Centers of America, Hollywood, Florida
  - Segal Institute For Clinical Research - West Broward Outpatient Clinic, Miami Lakes, Florida
  - Atlanta Center for Medical Research - Atlanta, Atlanta, Georgia
  - CBH Health, Gaithersburg, Maryland
  - St. Louis Clinical Trials, St Louis, Missouri
  - Altea Research Institute - Las Vegas, Las Vegas, Nevada
  - Hassman Research Institute, Marlton, New Jersey
  - Midwest Clinical Research Center, Dayton, Ohio
  - Carolina Clinical Trials, Charleston, South Carolina
  - Community Clinical Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Citrome L, Such P, Yildirim M, Madera-McDonough J, Beckham C, Zhang Z, Larsen F, Harlin M. Safety and Efficacy of Aripiprazole 2-Month Ready-to-Use 960 mg: Secondary Analysis of Outcomes in Adult Patients With Schizophrenia in a Randomized, Open-label, Parallel-Arm, Pivotal Study. J Clin Psychiatry. 2023 Sep 4;84(5):23m14873. doi: 10.4088/JCP.23m14873. PMID 37672016
- [Derived] McIntyre RS, Such P, Yildirim M, Madera-McDonough J, Zhang Z, Larsen F, Harlin M. Safety and efficacy of aripiprazole 2-month ready-to-use 960 mg: secondary analysis of outcomes in adult patients with bipolar I disorder in a randomized, open-label, parallel-arm, pivotal study. Curr Med Res Opin. 2023 Jul;39(7):1021-1030. doi: 10.1080/03007995.2023.2219155. Epub 2023 Jun 9. PMID 37272079
- [Derived] Harlin M, Yildirim M, Such P, Madera-McDonough J, Jan M, Jin N, Watkin S, Larsen F. A Randomized, Open-Label, Multiple-Dose, Parallel-Arm, Pivotal Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Aripiprazole 2-Month Long-Acting Injectable in Adults With Schizophrenia or Bipolar I Disorder. CNS Drugs. 2023 Apr;37(4):337-350. doi: 10.1007/s40263-023-00996-8. Epub 2023 Mar 24. PMID 36961650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 16 investigational sites in the United States from 01 August 2019 to 08 July 2020.
Groups:
- Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder: Participants with schizophrenia or bipolar I disorder received aripiprazole intra-muscularly (IM) 400 mg, for a total of 8 injections administered every 28 days (± 2 days) over the course of 32 weeks.
Period: Overall Study
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Started | 132 | 134
Safety Sample (Safety sample included all randomized participants who received at least 1 dose of aripiprazole injection, regardless of any protocol violation.) | 132 | 134
Efficacy Sample (Efficacy sample included all randomized participants who received at least 1 dose of aripiprazole injection and had at least 1 efficacy assessment.) | 132 | 134
Completed | 102 | 92
Not Completed | 30 | 42
Not completed — Adverse Event | 5 | 10
Not completed — Lost to Follow-up | 3 | 7
Not completed — Protocol Deviation | 2 | 2
Not completed — Withdrawal by Subject | 16 | 18
Not completed — Physician Decision | 1 | 1
Not completed — Due to Covid-19 | 2 | 3
Not completed — Not Due to Covid-19 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized sample consisted of all participants who were randomized.
Groups:
- Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder: Participants with schizophrenia or bipolar I disorder received aripiprazole 2M LAI 960 mg, for a total of 4 injections administered every 56 days (± 2 days) over the course of 32 weeks.
- Total: Total of all reporting groups
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder | Total
Number analyzed (Participants) | 132 | 134 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (10.8) | 46.8 (11.7) | 47.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 48 | 90
  Male | 90 | 86 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 119 | 122 | 241
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 29 | 33 | 62
  Race: Black or African American | 99 | 95 | 194
  Race: Asian | 3 | 4 | 7
  Race: Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. A TEAE is defined as an AE that started after investigational medicinal product (IMP) treatment; or if the event was continuous from baseline and was serious, IMP-related, or resulted in death, discontinuation, interruption, or reduction of the IMP.
Time Frame: From first dose of study drug up to 56 days (2M LAI 960 mg) or 28 days (IM depot 400 mg) post last dose of study drug (up to approximately 11 months)
Population: Safety sample included all randomized participants who received at least 1 dose of aripiprazole injection, regardless of any protocol violation.
Measure: Count of Participants; unit: Participants
Groups:
- Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder: Participants with schizophrenia or bipolar I disorder received aripiprazole 2M LAI 960 mg for a total of 4 injections administered every 56 days (± 2 days) over the course of 32 weeks.
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 132 | 134
Participants | 94 | 95

2. Primary Outcome: Number of Participants With Potentially Clinically Relevant Vital Signs Abnormalities
Description: Potentially clinically significant vital sign abnormalities included: heart rate supine (high: >120 beats per minute [BPM] and increase >=15 BPM; low: <50 BPM and decrease >=15 BPM), systolic blood pressure supine (high >180 (millimetres of mercury [mmHg] and increase >=20 mmHg); low: <90 mmHg and decrease >=20 mmHg), diastolic blood pressure supine (high: >105 mmHg and increase >=15 mmHg; low: <50 mmHg and decrease >=15 mmHg), heart rate standing (high: >120 BPM and increase >=15 BPM), systolic blood pressure standing (high: >180 mmHg and increase >= 20 mmHg; low: <90 mmHg and decrease >=20 mmHg), diastolic blood pressure standing (high: >105 mmHg and increase >=15 mmHg), weight in kilograms (kg) (high: increase >=7%; low: decrease >=7%), temperature (high: >=37.8 degree celsius [°C] and increase >=1.1°C), orthostatic hypotension (low: >=20 mmHg decrease in systolic blood pressure and >=25 BPM increase in heart rate from supine to standing.
Time Frame: From first dose of study drug up to Day 225
Population: Safety sample included all randomized participants who receive at least 1 dose of aripiprazole injection, regardless of any protocol violation. Overall number analyzed is the number of participants with data available for outcome measure analysis. 'Number Analyzed' signifies number of participants with data available for analysis of specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 131 | 133
Participants
  Heart Rate Supine: Low | 0 | 1
  Heart Rate Supine: High | 2 | 1
  Systolic Blood Pressure Supine: Low | 1 | 2
  Systolic Blood Pressure Supine: High | 0 | 1
  Diastolic Blood Pressure Supine: Low | 1 | 1
  Diastolic Blood Pressure Supine: High | 1 | 1
  Heart Rate Standing: High | 4 | 6
  Systolic Blood Pressure Standing: Low | 1 | 4
  Systolic Blood Pressure Standing: High | 0 | 2
  Diastolic Blood Pressure Standing: High | 2 | 3
  Weight: Low: number analyzed (Participants) | 128 | 126
  Weight: Low | 12 | 11
  Weight: High: number analyzed (Participants) | 128 | 126
  Weight: High | 52 | 54
  Temperature: High | 4 | 4
  Orthostatic Hypotension: Low | 2 | 2

3. Primary Outcome: Number of Participants With Potentially Clinically Relevant Electrocardiogram (ECG) Abnormalities
Description: Potentially clinically significant ECG abnormalities included rate: bradycardia (vent <=50 BPM] and decrease >=15 BPM); rhythm: sinus bradycardia (<= 50 BPM and decrease >= 15 BPM and no current diagnosis of atrial fibrillation, atrial flutter, or other rhythm abnormality); supraventricular premature beat (not present at baseline and present post baseline); ventricular premature beat (not present at baseline and present post baseline); conduction: right bundle branch block (not present at baseline and present post baseline); ST/T morphology: myocardial ischemia and symmetrical T-wave inversion (not present at baseline and present post baseline), QTcB, QTcF, and QTcN (>=450 milliseconds [msec] and >= 10% increase).
Time Frame: From first dose of study drug up to Day 225
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 130 | 131
Participants
  Bradycardia | 0 | 2
  Sinus Bradycardia | 0 | 2
  Supraventricular Premature Beat | 13 | 10
  Ventricular Premature Beat | 17 | 12
  Right Bundle Branch Block | 1 | 0
  Myocardial Ischemia | 3 | 7
  Symmetrical T-Wave Inversion | 12 | 12
  QTcB | 1 | 1
  QTcF | 0 | 1
  QTcN | 0 | 1

4. Primary Outcome: Number of Participants With Potentially Clinically Relevant Clinical Laboratory Abnormalities
Description: Potentially clinically relevant laboratory abnormalities included: In units per liter [U/L] (alanine aminotransferase: male[M]/female[F] >=3 x upper limit of normal (ULN); aspartate aminotransferase: M/F >= 3 x ULN; creatine kinase: M/F >= 3 x ULN); in milligrams per deciliter (mg/dL) (creatinine: M/F >= 2.0; glucose: M/F >= 200; urate: M >=10.5, F >=8.5); potassium [milliequivalents per liter (mEq/L)]: M/F >=5.5, in percentage (%) (eosinophils/leukocytes: M/F>=10%, hematocrit: M<=37%/F<=32% and 3 point decrease from baseline); hemoglobin (grams per deciliter [g/dL]): M<=11.5/F<=9.5; leukocytes [10^9 per liter (/L)]: M/F<=2.8 x 10^3 per microliters (/uL); platelets (10^9/L): M/F>=700 x 10^3/uL; glucose, urine and protein, urine: increase of >=2 units; and prolactin (nanograms per milliliter [ng/mL]: M/F > 1 x ULN.
Time Frame: From first dose of study drug up to Day 225
Population: Safety sample included all randomized participants who received at least 1 dose of aripiprazole injection, regardless of any protocol violation. Overall number analyzed is the number of participants with data available for outcome measure analysis. 'Number Analyzed' signifies number of participants with data available for analysis of specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 129 | 126
Participants
  High Alanine Aminotransferase (U/L): number analyzed (Participants) | 128 | 126
  High Alanine Aminotransferase (U/L) | 1 | 2
  High Aspartate Aminotransferase (U/L): number analyzed (Participants) | 128 | 126
  High Aspartate Aminotransferase (U/L) | 0 | 2
  High Creatine Kinase (U/L): number analyzed (Participants) | 128 | 126
  High Creatine Kinase (U/L) | 12 | 1
  High Creatinine (mg/dL): number analyzed (Participants) | 128 | 126
  High Creatinine (mg/dL) | 2 | 1
  High Glucose (mg/dL): number analyzed (Participants) | 128 | 126
  High Glucose (mg/dL) | 7 | 3
  High Potassium (mEq/L): number analyzed (Participants) | 128 | 126
  High Potassium (mEq/L) | 5 | 4
  High Urate (mg/dL): number analyzed (Participants) | 128 | 126
  High Urate (mg/dL) | 2 | 0
  High Eosinophils/Leukocytes (%) | 2 | 0
  Low Hematocrit (%) | 7 | 8
  Low Hemoglobin (g/dL) | 4 | 9
  Low Leukocytes (10^9/L) | 0 | 3
  High Platelets (10^9/L) | 0 | 1
  High Glucose, Urine: number analyzed (Participants) | 128 | 126
  High Glucose, Urine | 5 | 6
  High Protein, Urine: number analyzed (Participants) | 128 | 126
  High Protein, Urine | 1 | 2
  High Prolactin (ng/mL): number analyzed (Participants) | 123 | 118
  High Prolactin (ng/mL) | 2 | 4

5. Primary Outcome: Mean Change From Baseline in Simpson-Angus Neurologic Rating Scale (SAS) Total Score
Description: The SAS scale is used to evaluate extrapyramidal symptoms (EPS) and consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item is rated on a 5-point scale, with a score of range of 0 (absence of symptoms) to 4 (severe condition). The SAS total score is the sum of the scores for all 10 items, possible total score is 0 to 40. Negative change from baseline indicates less symptoms.
Time Frame: Baseline, Week 32
Population: Safety sample included all randomized participants who received at least 1 dose of aripiprazole injection, regardless of any protocol violation. 'Number Analyzed' signifies number of participants with available data for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 132 | 134
score on a scale
  Baseline | 0.2 (0.6) | 0.2 (0.4)
  Change From Baseline at Week 32: number analyzed (Participants) | 131 | 133
  Change From Baseline at Week 32 | -0.0 (0.7) | 0.1 (0.6)

6. Primary Outcome: Mean Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Movement Score
Description: The AIMS assessment consists of 10 items describing symptoms of dyskinesia. Facial and oral movements (items 1 through 4), extremity movements (items 5 and 6), and trunk movements (item 7), dyskinesias (items 8 through 10). Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms (for item 10, no awareness), and a score of 4 indicating a severe condition (for item 10, aware/severe distress). AIMS movement score is the sum of the ratings for the first seven items with the possible total scores of 0 to 28. Negative change from baseline indicates less symptoms.
Time Frame: Baseline, Week 32
Population: Safety sample included all randomized participants who receive at least 1 dose of aripiprazole injection, regardless of any protocol violation. 'Number Analyzed' signifies number of participants with available data for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 132 | 134
score on a scale
  Baseline | 0.1 (1.0) | 0.1 (0.7)
  Change from Baseline at Week 32: number analyzed (Participants) | 131 | 133
  Change from Baseline at Week 32 | 0.0 (0.5) | -0.1 (0.6)

7. Primary Outcome: Mean Change From Baseline in Barnes Akathisia Rating Score (BARS) Global Score
Description: The BARS consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the participant, participant distress due to akathisia, and global evaluation of akathisia. The first 3 items are rated on a 4-point scale, with a score of 0 representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation is made on a 6-point scale, with 0 representing absence of symptoms and a score of 5 representing severe akathisia. Total BARS score ranges from 0 to 14 where lower scores indicate less symptoms and negative change from baseline indicate less symptoms.
Time Frame: Baseline, Week 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 132 | 134
score on a scale
  Baseline | 0.1 (0.3) | 0.1 (0.3)
  Change from Baseline at Week 32: number analyzed (Participants) | 131 | 133
  Change from Baseline at Week 32 | 0.1 (0.6) | 0.1 (0.4)

8. Primary Outcome: Visual Analog Scale (VAS) Scores for Pain Perception of Aripiprazole 2M LAI 960 mg
Description: Injection-site pain was evaluated by mean VAS scores as reported by the participant after each injection at visits where an injection occurred. The last injection was the final injection for any given participant. Ratings ranged from 0 (no pain) to 100 (unbearably painful).
Time Frame: Day 1 (First injection) to Day 169 (Last injection)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 132
score on a scale
  First Injection: Predose: number analyzed (Participants) | 131
  First Injection: Predose | 1.0 (1.29)
  First Injection: Post dose: number analyzed (Participants) | 130
  First Injection: Post dose | 3.7 (9.09)
  Second Injection: Predose: number analyzed (Participants) | 113
  Second Injection: Predose | 1.0 (2.32)
  Second Injection: Post dose: number analyzed (Participants) | 113
  Second Injection: Post dose | 1.4 (2.78)
  Third Injection: Predose: number analyzed (Participants) | 109
  Third Injection: Predose | 1.0 (2.58)
  Third Injection: Post dose: number analyzed (Participants) | 105
  Third Injection: Post dose | 2.0 (6.01)
  Fourth Injection: Predose: number analyzed (Participants) | 103
  Fourth Injection: Predose | 0.8 (1.02)
  Fourth Injection: Post dose: number analyzed (Participants) | 102
  Fourth Injection: Post dose | 1.4 (4.38)
  Last Injection: Predose | 0.8 (1.03)
  Last Injection: Post dose: number analyzed (Participants) | 130
  Last Injection: Post dose | 1.4 (3.98)

9. Primary Outcome: VAS Scores for Pain Perception of Aripiprazole IM Depot 400 mg
Description: as for outcome 8
Time Frame: Day 1 (First injection) to Day 197 (Last injection)
Population: Safety sample included all randomized participants who receive at least 1 dose of aripiprazole injection, regardless of any protocol violation. 'Number Analyzed' signifies number of participants with available data for this outcome measure at the specified timepoint. Participants whose VAS scores were analyzed for pain perception, are reported in this outcome measure, and may differ from participants who were assessed by Investigator for pain on 4-point scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 134
score on a scale
  First Injection: Predose | 1.6 (2.37)
  First Injection: Post dose: number analyzed (Participants) | 130
  First Injection: Post dose | 3.0 (5.28)
  Second Injection: Predose: number analyzed (Participants) | 117
  Second Injection: Predose | 1.5 (2.66)
  Second Injection: Post dose: number analyzed (Participants) | 112
  Second Injection: Post dose | 1.6 (3.09)
  Third Injection: Predose: number analyzed (Participants) | 107
  Third Injection: Predose | 0.8 (1.10)
  Third Injection: Post dose: number analyzed (Participants) | 103
  Third Injection: Post dose | 1.2 (2.09)
  Fourth Injection: Predose: number analyzed (Participants) | 103
  Fourth Injection: Predose | 0.7 (0.79)
  Fourth Injection: Post dose: number analyzed (Participants) | 102
  Fourth Injection: Post dose | 1.1 (2.39)
  Fifth Injection: Predose: number analyzed (Participants) | 99
  Fifth Injection: Predose | 0.7 (0.82)
  Fifth Injection: Post dose: number analyzed (Participants) | 99
  Fifth Injection: Post dose | 0.8 (1.12)
  Sixth Injection: Predose: number analyzed (Participants) | 97
  Sixth Injection: Predose | 0.8 (1.11)
  Sixth Injection: Post dose: number analyzed (Participants) | 96
  Sixth Injection: Post dose | 0.8 (1.20)
  Seventh Injection: Predose: number analyzed (Participants) | 92
  Seventh Injection: Predose | 0.6 (0.77)
  Seventh Injection: Post dose: number analyzed (Participants) | 90
  Seventh Injection: Post dose | 1.0 (2.30)
  Eighth Injection: Predose: number analyzed (Participants) | 89
  Eighth Injection: Predose | 0.6 (0.69)
  Eighth Injection: Post dose: number analyzed (Participants) | 89
  Eighth Injection: Post dose | 0.8 (0.85)
  Last Injection: Predose: number analyzed (Participants) | 132
  Last Injection: Predose | 0.9 (1.00)
  Last Injection: Post dose: number analyzed (Participants) | 131
  Last Injection: Post dose | 1.3 (2.62)

10. Primary Outcome: Number of Participants With Injection Site Evaluations (Pain, Redness, Swelling, Induration) Measured by Investigator Rating After Aripiprazole 2M LAI 960 mg Injection
Description: Injection-site reactions were assessed by the investigator (or qualified designee) and the participant. Investigators rated localized pain, redness, swelling, and induration at the most recent injection site using a 4-point categorical scale (absent, mild, moderate, severe). The participant indicated the degree of pain at the most recent injection site using a VAS instrument. Ratings included were: 0 = absent, 1 = mild, 2 = moderate, 3 = severe. The last injection was the final injection for any given participant.
Time Frame: Day 1 (First injection) to Day 169 (Last injection)
Population: Safety sample included all randomized participants who received at least 1 dose of aripiprazole injection, regardless of any protocol violation. Overall number analyzed is the number of participants with data available for outcome measure analysis. 'Number Analyzed' signifies number of participants with available data for this outcome measure at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 131
Participants
  First Injection: Mild Pain: number analyzed (Participants) | 130
  First Injection: Mild Pain | 11
  Second Injection: Mild Pain: number analyzed (Participants) | 114
  Second Injection: Mild Pain | 2
  Third Injection: Mild Pain: number analyzed (Participants) | 108
  Third Injection: Mild Pain | 5
  Fourth Injection: Mild Pain: number analyzed (Participants) | 102
  Fourth Injection: Mild Pain | 5
  Last injection: Mild Pain | 5
  First injection: Mild Redness: number analyzed (Participants) | 130
  First injection: Mild Redness | 3
  Third injection: Mild Redness: number analyzed (Participants) | 108
  Third injection: Mild Redness | 1
  Last injection: Mild Redness | 1

11. Primary Outcome: Number of Participants With Injection Site Evaluations (Pain, Redness, Swelling, Induration) Measured by Investigator Rating After Aripiprazole IM Depot 400 mg Injection
Description: as for outcome 10
Time Frame: Day 1 (First injection) to Day 197 (Last injection)
Population: Safety sample included all randomized participants who received at least 1 dose of aripiprazole injection, regardless of any protocol violation. 'Number Analyzed' signifies number of participants with available data for this outcome measure at the specified timepoint. Participants whose injection-site reactions were assessed by the investigator, are reported in this outcome measure, and may differ from participants whose VAS scores were assessed for pain.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 134
Participants
  First Injection: Mild Pain: number analyzed (Participants) | 131
  First Injection: Mild Pain | 7
  Second Injection: Mild Pain: number analyzed (Participants) | 116
  Second Injection: Mild Pain | 3
  Third Injection: Mild Pain: number analyzed (Participants) | 109
  Third Injection: Mild Pain | 7
  Fourth Injection: Mild Pain: number analyzed (Participants) | 105
  Fourth Injection: Mild Pain | 1
  Fifth Injection: Mild Pain: number analyzed (Participants) | 101
  Fifth Injection: Mild Pain | 3
  Seventh Injection: Mild Pain: number analyzed (Participants) | 94
  Seventh Injection: Mild Pain | 1
  Eighth Injection: Mild Pain: number analyzed (Participants) | 90
  Eighth Injection: Mild Pain | 1
  Last injection: Mild Pain | 3
  First injection: Mild Redness: number analyzed (Participants) | 132
  First injection: Mild Redness | 1
  Second injection: Mild Redness: number analyzed (Participants) | 116
  Second injection: Mild Redness | 3

12. Primary Outcome: Number of Participants With Suicidality as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS was used to assess the suicidality of participants during the study. The assessment included "yes" or "no" responses for 5 questions, each related to suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Numeric ratings were provided for suicidal ideation: Score range of 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent), higher total scores indicate more suicidal ideation; Suicidal behavior: Score range of 0 (no suicidal behavior) to 4 (actual suicide attempt), higher total scores indicate more suicidal behavior. Suicidality was defined as reporting any suicidal ideation or behavior.
Time Frame: Baseline to Day 225
Population: Safety sample included all randomized participants who received at least 1 dose of aripiprazole injection, regardless of any protocol violation. Overall number analyzed is the number of participants with data available for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 130 | 132
Participants | 4 | 4

13. Primary Outcome: Plasma Concentration of Aripiprazole 56 Days Postdose (C56) of Aripiprazole 2M LAI 960 mg After the Fourth Dose
Time Frame: Day 225
Population: Pharmacokinetics (PK) sample included all dosed participants who had 1 or more evaluable aripiprazole PK parameters. Overall number analyzed is the number of participants with data available for outcome measure (OM) analysis. As pre-specified in protocol and SAP, data for this OM was reported for participants with schizophrenia or bipolar I disorder who received aripiprazole 2M LAI 960 mg.
Measure: Mean (Standard Deviation); unit: ng/mL (nanogram per milliliter)
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 96
ng/mL (nanogram per milliliter) | 250 (128)

14. Primary Outcome: Plasma Concentration of Aripiprazole 28 Days Postdose (C28) of Aripiprazole IM Depot 400 mg After the Eighth Dose
Time Frame: Day 225
Population: PK sample included all dosed participants who had 1 or more evaluable aripiprazole PK parameters. Overall number analyzed is the number of participants with data available for outcome measure analysis. As pre-specified in protocol and SAP, data for this OM was reported for participants with schizophrenia or bipolar I disorder who received aripiprazole IM Depot 400 mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 82
ng/mL | 257 (162)

15. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 28 Days (AUC0-28) of Aripiprazole After the Seventh and Eighth Doses of Aripiprazole IM Depot 400 mg
Time Frame: Days 169 (predose and 4, 8, 12 hours post dose), 170, 171, 173, 176, 178, 181, 183, 186, 190, 197 (predose and 4, 8, 12 hours post dose), 198, 199, 201, 204, 206, 209, 211, 214, 218, 225
Population: PK sample included all dosed participants who had 1 or more evaluable aripiprazole PK parameters. Overall number analyzed is the number of participants with data available for outcome measure analysis. 'Number Analyzed' signifies number of participants with available data for this outcome measure at the specified timepoint. As pre-specified in protocol and SAP, data for this OM was reported for participants with schizophrenia or bipolar I disorder who received aripiprazole IM Depot 400 mg.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 33
day*ng/mL
  AUC0-28 After Seventh Dose (Day 169) | 7760 (4300)
  AUC0-28 After Eighth Dose (Day 197): number analyzed (Participants) | 32
  AUC0-28 After Eighth Dose (Day 197) | 7840 (5170)

16. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 56 Days (AUC0-56) of Aripiprazole After the Fourth Dose of Aripiprazole 2M LAI 960 mg
Time Frame: Days 169 (predose and 4, 8, 12 hours post dose), 170, 171, 173, 176, 178, 181, 183, 186, 190, 197, 204, 211, 218, and 225
Population: PK sample included all dosed participants who had 1 or more evaluable aripiprazole PK parameters. Overall number analyzed is the number of participants with data available for outcome measure analysis. As pre-specified in protocol and SAP, data for this OM was reported for participants with schizophrenia or bipolar I disorder who received aripiprazole 2M LAI 960 mg.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 34
day*ng/mL | 14700 (7460)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Aripiprazole After First and Fourth Doses of Aripiprazole 2M LAI 960 mg
Time Frame: Days 1(predose [within 2 hours(h) prior to dosing]&4,8,12 h postdose),2,3,5,8,10,13,15,18,22,29,36,43,50,57(predose),85,113(predose),141,169(predose [within 2 h prior to dosing]& 4,8,12 h postdose),170,171,173,176,178,181,183,186,190,197,204,211,218 & 225
Population: PK sample included all dosed participants who have 1 or more evaluable aripiprazole PK parameters. Overall number analyzed is the number of participants with data available for outcome measure analysis. 'Number Analyzed' signifies number of participants with available data for this outcome measure at the specified timepoint. As pre-specified in protocol and SAP, data for this OM was reported for participants with schizophrenia or bipolar I disorder who received aripiprazole 2M LAI 960 mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 37
ng/mL
  Cmax After First Dose (Day 1) | 286 (203)
  Cmax After Fourth Dose (Day 169): number analyzed (Participants) | 34
  Cmax After Fourth Dose (Day 169) | 342 (157)

18. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Aripiprazole After First and Fourth Doses of Aripiprazole 2M LAI 960 mg
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: days
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 37
days
  Tmax After First Dose (Day 1) | 8.58 [3.92 to 55.9]
  Tmax After Fourth Dose (Day 169): number analyzed (Participants) | 34
  Tmax After Fourth Dose (Day 169) | 28.0 [0.930 to 49.0]

19. Secondary Outcome: AUC0-56 After the First Dose of Aripiprazole 2M LAI 960 mg
Time Frame: Days 1 (predose and 4, 8, 12 hours post-dose), 2, 3, 5, 8, 10, 13, 15, 18, 22, 29, 36, 43, 50 and 57 (pre-dose)
Population: PK sample included all dosed participants who have 1 or more evaluable aripiprazole PK parameters. Overall number analyzed is the number of participants with data available for outcome measure analysis. As pre-specified in protocol and SAP, data for this OM was reported for participants with schizophrenia or bipolar I disorder who received aripiprazole 2M LAI 960 mg.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 37
day*ng/mL | 9180 (4940)

20. Secondary Outcome: Plasma Concentration of Aripiprazole 56 Days (C56) After the First Dose of Aripiprazole 2M LAI 960 mg
Time Frame: Predose on Day 57
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 113
ng/mL | 165 (91.7)

21. Secondary Outcome: AUC0-28 After the Fourth Dose of Aripiprazole 2M LAI 960 mg
Time Frame: Days 169 (predose and 4, 8, 12 hours postdose), 170, 171, 173, 176, 178, 181, 183, 186, 190, and 197
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 34
day*ng/mL | 7190 (3470)

22. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 29 to 56 Days (AUC29-56) After the Fourth Dose of Aripiprazole 2M LAI 960 mg
Time Frame: Days 204, 211, 218, and 225
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 34
day*ng/mL | 7500 (4200)

23. Secondary Outcome: Peak-to-Trough Percent Fluctuation (PTF%) After the Fourth Dose of Aripiprazole 2M LAI 960 mg
Description: PTF% was determined as 100*(Cmax - Cmin [minimum plasma concentration of the drug])/Caverage (average steady-state plasma drug concentration during multiple-dose administration) following fourth dose.
Time Frame: Days 169 (Predose [within 2 hours prior to dosing] and 4, 8, 12 hours post dose), 170, 171, 173, 176, 178, 181, 183, 186, 190, 197, 204, 211, 218, and 225
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage fluctuation
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 34
percentage fluctuation | 63.4 (25.1)

24. Secondary Outcome: Cmax of Aripiprazole After the First, Seventh, and Eighth Doses of Aripiprazole IM Depot 400 mg
Time Frame: Predose [within 2 hours prior to dosing; 4,8,12h postdose] on Days 1,169,197; Predose on Days 29,57,85,113,141; and on Days 2, 3, 5, 8, 10, 13, 15, 18, 22, 170, 171, 173, 176, 178, 181, 183, 186, 190,198, 199, 201, 204, 206, 209, 211, 214, 218, 225
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 35
ng/mL
  Cmax After First Dose (Day 1) | 280 (123)
  Cmax After Seventh Dose (Day 169): number analyzed (Participants) | 33
  Cmax After Seventh Dose (Day 169) | 339 (168)
  Cmax After Eighth Dose (Day 197): number analyzed (Participants) | 32
  Cmax After Eighth Dose (Day 197) | 344 (212)

25. Secondary Outcome: Tmax of Aripiprazole After the First, Seventh, and Eighth Doses of Aripiprazole IM Depot 400 mg
Time Frame: as for outcome 24
Population: as for outcome 15
Measure: Median (Full Range); unit: days
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 35
days
  Tmax After First Dose (Day 1) | 9.04 [3.83 to 27.9]
  Tmax After Seventh Dose (Day 169): number analyzed (Participants) | 34
  Tmax After Seventh Dose (Day 169) | 6.97 [1.05 to 28.0]
  Tmax After Eighth Dose (Day 197): number analyzed (Participants) | 34
  Tmax After Eighth Dose (Day 197) | 4.07 [0 to 28.0]

26. Secondary Outcome: AUC0-28 After the First Dose of Aripiprazole IM Depot 400 mg
Time Frame: Days 1 (predose and 4, 8, and 12 hours postdose), 2, 3, 5, 8, 10, 13, 15, 18, 22 and 29 (predose)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 35
day*ng/mL | 5030 (2580)

27. Secondary Outcome: Plasma Concentration of Aripiprazole 28 Days (C28) After the First Dose of Aripiprazole IM Depot 400 mg
Time Frame: Predose on Day 29
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 110
ng/mL | 112 (82.9)

28. Secondary Outcome: PTF% After the Eighth Dose of Aripiprazole IM Depot 400 mg
Description: PTF% was determined as 100*(Cmax - Cmin [minimum plasma concentration of the drug])/Caverage (average steady-state plasma drug concentration during multiple-dose administration) following eighth dose.
Time Frame: Days 197 (Predose [within 2 hours prior to dosing] and 4, 8, 12 hours post dose),198, 199, 201, 204, 206, 209, 211, 214, 218, 225
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage fluctuation
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 34
percentage fluctuation | 48.3 (19.0)

29. Secondary Outcome: Plasma Concentration of Aripiprazole 7 Days Post First Dose (C7) of Aripiprazole 2M LAI 960 mg
Time Frame: Day 8
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 41
ng/mL | 221 (178)

30. Secondary Outcome: Plasma Concentration of Aripiprazole Post First Dose (C14) of Aripiprazole IM Depot 400 mg
Time Frame: Day 15
Population: PK sample included all dosed participants who have 1 or more evaluable aripiprazole PK parameters. Overall number analyzed is the number of participants with data available for outcome measure analysis. As pre-specified in protocol and SAP, data for this OM was reported for participants with schizophrenia or bipolar I disorder who received aripiprazole IM Depot 400 mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 39
ng/mL | 229 (121)

31. Secondary Outcome: Mean Change From Baseline in Positive and Negative Syndrome Scale Rating Criteria (PANSS) Total Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome). Higher scores indicate worse condition. The PANSS was assessed for schizophrenia participants only.
Time Frame: Baseline, Week 32
Population: Efficacy sample set included all randomized participants who received at least 1 dose of aripiprazole injection and have had at least 1 efficacy assessment. Overall number analyzed is the number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aripiprazole 2M LAI 960 mg: Schizophrenia: Participants with schizophrenia received aripiprazole 2M LAI 960 mg, for a total of 4 injections administered every 56 days (± 2 days) over the course of 32 weeks.
- Aripiprazole IM Depot 400 mg: Schizophrenia: Participants with schizophrenia received aripiprazole IM 400 mg, for a total of 8 injections administered every 28 days (± 2 days) over the course of 32 weeks.
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia | Aripiprazole IM Depot 400 mg: Schizophrenia
Number analyzed (Participants) | 89 | 85
score on a scale | -2.6 (11.7) | -1.7 (8.5)

32. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression - Severity Scale (CGI-S) Score
Description: The CGI-S is a standardized, clinician-administered global rating scale that measures disease severity. To assess CGI-S, the rater or investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices include: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. The cumulative score range is 0-7. A higher score on the CGI-S represents a higher severity of disease. The CGI-S scale was assessed for schizophrenia participants only.
Time Frame: Baseline, Week 32
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia | Aripiprazole IM Depot 400 mg: Schizophrenia
Number analyzed (Participants) | 89 | 85
score on a scale | -0.3 (0.6) | -0.1 (0.7)

33. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression - Improvement Scale (CGI-I) Score
Description: The CGI-I scale is a clinician rated scale which assesses the improvement of illness for each participant. To assess CGI-I, the rater or investigator rated the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared with the participant's condition at baseline. Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Scores range from 0 to 7. Higher scores indicate worse condition.
Time Frame: Baseline, Week 32
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 123 | 117
score on a scale | 3.4 (1.1) | 3.5 (1.1)

34. Secondary Outcome: Mean Change From Baseline in Subjective Well-Being Under Neuroleptic Treatment-Short Form (SWN-S) Total Score
Description: The participant's feeling of their own well-being was assessed using the 20-question SWN-S. The SWN-S was a validated self-report instrument that evaluated the participant's perception of well-being while receiving antipsychotic medication. The questionnaire consisted of 20 items (10 positive and 10 negative statements) and 5 subscales (mental functioning, social integration, emotional regulation, physical functioning, self-control) whose items followed in random order. For items marked with a '+', the response choices and scoring is not at all = 1, hardly at all = 2, a little = 3, somewhat = 4, much = 5, and very much = 6. For items marked with a '- ', the scoring is reversed; response choices and scoring are as follows: not at all = 6, hardly at all = 5, a little = 4, somewhat = 3, much = 2, very much = 1. SWN-S subscale score's each item was rated on a score of 1 (none) to 6 (severe), and total score ranged from 20 to 120, with higher scores indicating stronger subjective feeling
Time Frame: Baseline, Week 32
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
Number analyzed (Participants) | 125 | 121
score on a scale | 3.2 (15.8) | 0.5 (18.2)

35. Secondary Outcome: Mean Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a diagnostic questionnaire used by clinician to assess the participant's severity of depression. This scale consists of 10 items each with 7 defined grades of severity on 0 to 6 scale (reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). MADRS total score is sum of 10 individual item scores ranging from 0-60 categorized as: 0 to 6: normal/symptoms absent, 7 to 19: mild depression, 20 to 34: moderate depression, and 35 to 60: severe depression. Higher score indicates more depressive symptoms. The MADRS was assessed for bipolar I disorder participants only.
Time Frame: Baseline, Week 32
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aripiprazole 2M LAI 960 mg: Bipolar I Disorder: Participants with bipolar I disorder received aripiprazole 2M LAI 960 mg, for a total of 4 injections administered every 56 days (± 2 days) over the course of 32 weeks.
- Aripiprazole IM Depot 400 mg: Bipolar I Disorder: Participants with bipolar I disorder received aripiprazole IM 400 mg, for a total of 8 injections administered every 28 days (± 2 days) over the course of 32 weeks.
Arm/Group | Aripiprazole 2M LAI 960 mg: Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Bipolar I Disorder
Number analyzed (Participants) | 39 | 40
score on a scale | -3.5 (9.1) | -3.3 (12.5)

36. Secondary Outcome: Mean Change From Baseline in Young Mania Rating Scale (YMRS) Total Score
Description: The YMRS is an 11-item, multiple-choice diagnostic questionnaire which psychiatrists use to assess the core symptoms of mania and is based on the participants subjective report of their condition. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Total score is summed of 11 items. Total score range is from 0 to 60 and the higher score represent a worse outcome. The YMRS was assessed for bipolar I disorder participants only.
Time Frame: Baseline, Week 32
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Bipolar I Disorder
Number analyzed (Participants) | 39 | 40
score on a scale | -1.9 (7.1) | -4.7 (7.7)

37. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression - Bipolar Version (CGI-BP) Severity of Illness Score
Description: The CGI-BP scale refers to the global impression of the participants with respect to bipolar disorder. The scale rates the participant's severity of illness (CGI-BP-Severity: mania, depression, and overall bipolar illness) and change from preceding phase (CGI-BP change from preceding phase: mania, depression, and overall bipolar illness) based on a 7-point scale ranging from 1 (normal, not ill) to 7 (very severely ill). A negative change score signifies improvement. The CGI-BP was assessed for bipolar I disorder participants only.
Time Frame: Baseline, Week 32
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole 2M LAI 960 mg: Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Bipolar I Disorder
Number analyzed (Participants) | 39 | 40
score on a scale | -0.2 (1.0) | -0.6 (1.2)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 56 days (2M LAI 960 mg) or 28 days (IM depot 400 mg) post last dose of study drug (up to approximately 11 months)
Description: Safety sample included all randomized participants who received at least 1 dose of aripiprazole injection, regardless of any protocol violation.
Arm/Group | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder
All-Cause Mortality (participants affected / at risk) | 1/132 | 0/134
Serious Adverse Events (participants affected / at risk) | 6/132 | 8/134
Other Adverse Events (participants affected / at risk) | 92/132 | 92/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder (N=132) | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder (N=134)
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Akathisia (Nervous system disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Depressive Symptom (Psychiatric disorders) | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 2 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 2M LAI 960 mg: Schizophrenia or Bipolar I Disorder (N=132) | Aripiprazole IM Depot 400 mg: Schizophrenia or Bipolar I Disorder (N=134)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 3 | 5
Constipation (Gastrointestinal disorders) | 8 | 8
Dental Caries (Gastrointestinal disorders) | 1 | 0
Dental Discomfort (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2
Gingival Swelling (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 2 | 10
Vomiting (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 3 | 2
Injection Site Discomfort (General disorders) | 1 | 0
Injection Site Mass (General disorders) | 1 | 0
Injection Site Pain (General disorders) | 24 | 12
Oedema Peripheral (General disorders) | 1 | 1
Bacterial Vaginosis (Infections and infestations) | 1 | 0
Body Tinea (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 2 | 1
Infected Bite (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Localised Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4
Periodontitis (Infections and infestations) | 0 | 1
Pustule (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 3 | 2
Tooth Abscess (Infections and infestations) | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 3
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 1
Burns First Degree (Injury, poisoning and procedural complications) | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 1
Nail Injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 3 | 2
Blood Pressure Increased (Investigations) | 1 | 2
Blood Prolactin Increased (Investigations) | 1 | 0
Blood Triglycerides Increased (Investigations) | 1 | 0
Body Temperature Increased (Investigations) | 1 | 0
Electrocardiogram T Wave Inversion (Investigations) | 0 | 1
Heart Rate Increased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1
Liver Function Test Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 2 | 3
Weight Increased (Investigations) | 30 | 28
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Akathisia (Nervous system disorders) | 13 | 12
Bradykinesia (Nervous system disorders) | 1 | 0
Disturbance In Attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dyskinesia (Nervous system disorders) | 4 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Extrapyramidal Disorder (Nervous system disorders) | 2 | 1
Head Titubation (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 10 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intention Tremor (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 1
Oromandibular Dystonia (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 6 | 4
Tension Headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 4
Agitation (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 11 | 10
Bipolar Disorder (Psychiatric disorders) | 2 | 0
Bruxism (Psychiatric disorders) | 1 | 0
Depressed Mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Depressive Symptom (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 10 | 11
Libido Decreased (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Psychotic Symptom (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 3 | 0
Schizophrenia (Psychiatric disorders) | 5 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 2 | 2
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/43/NCT04030143/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT04030143/SAP_001.pdf